CLINICAL TRIAL: NCT05958212
Title: The Efficacy of Unilateral Speed-upscaling Gait Training in Promoting Pain and Functional Recovery in People With Total Knee Replacement: A Randomised Controlled Trial
Brief Title: Innovative Gait Training for People With Knee Osteoarthritis Using Dual Belt Treadmill
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Hong Kong Buddhist Hospital (Unknown); The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Dr Patrick Kwong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0212
Record Dates: First submitted 2023-06-19; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive a weekly gait training program at PolyU in addition to conventional treatment at Outpatient Patient Department (OPD) of The Hong Kong Buddhist Hospital twice per week for 4 consecutive weeks. Gait training program at PolyU is a supervised rehabilitation program performed on the dual-belt treadmill.
  Interventions: Behavioral: Gait training program
- Control Group (Active Comparator): Participants in control group will only receive conventional treatment at Outpatient Patient Department (OPD) of BH twice per week for 4 consecutive weeks.
  Interventions: Behavioral: Conventional training only

INTERVENTIONS:
Behavioral: Gait training program — Gait training program at PolyU is a supervised rehabilitation program performed on the dual-belt treadmill. It consists of forward walking at increased speed over the affected leg and retro walking (backward walking) at individual's own pace (5 minutes/set for three sets, with rest periods in each session). This program also consists of a standardized set of warm-up and cool-down exercises at each training session.
  Participants will also receive conventional physiotherapy treatment in the outpatient physiotherapy clinic.
  Arms: Intervention Group
Behavioral: Conventional training only — Conventional physiotherapy treatment in the outpatient physiotherapy clinic.
  Arms: Control Group

SUMMARY:
Knee osteoarthritis (OA) is the most common form of arthritis and is the leading cause of chronic musculoskeletal pain and functional disability. Gait assessment is essential for the rehabilitation of people with knee OA. It may reflect the impact of knee OA on functional outcomes and allow prediction of prognosis for patients. Various people with knee OA may demonstrate different forms of gait asymmetry owing to his/her own knee pain experienced and joint instability perceived. The stance time, peak vertical and peak propulsive ground reaction force have found to be significantly reduced on the OA affected limb. People with knee OA demonstrate compensatory gait pattern to minimize joint loading. It is quite common that the severity of the OA symptoms varies in the two knees, and patients may demonstrate various forms of gait asymmetries, such changes in gait biomechanics does not only impact the affected knee joint. Its impact extends proximally along the kinetic chain system of the human body, where often knee OA patients presents with significantly increased lateral trunk flexion towards ipsilateral limb during walking.

Gait asymmetry as a result of knee OA has been constantly reported in both human and animal studies. Previous studies showed that people with unilateral knee symptoms may adapt to asymmetrical movement patterns, which results in reduced net knee extension demand moments Research interest on gait asymmetry has been expanded to other cohort of patients, e.g. hemiplegic stroke patients. Extensive evidence has shown that the modification of walking speed has a positive impact on the propulsive force of hemiplegic patient's affected limb. These encouraging results have form indications for future investigation on evaluating the impact of innovative gait training in promoting symmetrical gait pattern, targeting patients with unilateral knee OA or bilateral knee OA of different severity. The objective to assess knee OA's gait under different walking conditions is now feasible with the access to the dualbelt treadmill at PolyU. In addition to walking speed modification, emerging backward walking as part of gait training rehabilitation in knee OA patients has become increasingly popular. Backward walking is regulated by the same central pattern generator as forward walking; however, it does not require initial heel contact in early stance phase of the gait cycle as it would be in forward walking. This leads to reduced compression force at the patella-femoral joint and decreased force absorption imposed at the knee joint. Recent systematic review and meta-analysis have suggested combining backward walking to conventional physiotherapy has significantly improve clinical outcomes, including pain control, functional disability, muscle strength, gait pattern, balance and postural stability in knee OA patients.

All of above-mentioned findings have highlighted the connection between specific gait parameters and clinical outcomes, and also the importance of monitoring these changes as disease naturally progress. It is also vital to note the benefits of emerging technologies as the implementation of novel strategies can optimize the ambulatory capacity of the individual, which therefore enhance their recovery potential and quality of life.

DETAILED DESCRIPTION:
This study is a two-armed, parallel group, single centered randomized controlled trial investigating the efficacy of gait training combined with conventional treatment as compared to conventional treatment alone in post-TKR rehabilitation program. Potential participants will be recruited from BH and QEH, where patients with confirmed diagnosis of K&L grade 2 to 4 knee OA who have received TKR will be eligible for this study. Subjects with prior history of knee surgery, impaired lower limb function other than knee joint or has previously received an intra-articular injection to knee will be excluded from the study to ensure validity of results. It aims to compare and evaluate the effectiveness of combined conventional rehabilitation with gait training on dual-belt treadmill and conventional rehabilitation alone on post-operative clinical outcomes and gait pattern.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be recruited from BH and QEH, where patients with confirmed diagnosis of K&L grade 2 to 4 knee OA who have received TKR will be eligible for this study.

Exclusion Criteria:

* Subjects with prior history of knee surgery, impaired lower limb function other than knee joint or has previously received an intra-articular injection to knee will be excluded from the study to ensure validity of results.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index | pre-operative session (T1)
  Pain intensity, stiffness and function of the operated knee will be assessed using the Western Ontario and McMaster Universities Arthritis Index.
  Minimum：0 Maximum：96 Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster Universities Arthritis Index | two-weeks post-operation (T2)
  Pain intensity, stiffness and function of the operated knee will be assessed using the Western Ontario and McMaster Universities Arthritis Index.
  Minimum：0 Maximum：96 Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster Universities Arthritis Index | six-weeks post-operation(T3)
  Pain intensity, stiffness and function of the operated knee will be assessed using the Western Ontario and McMaster Universities Arthritis Index.
  Minimum：0 Maximum：96 Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster Universities Arthritis Index | six-month follow-up
  Pain intensity, stiffness and function of the operated knee will be assessed using the Western Ontario and McMaster Universities Arthritis Index.
  Minimum：0 Maximum：96 Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
30s Chair-Stand Test | pre-operative session (T1)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
30s Chair-Stand Test | two-weeks post-operation (T2)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
30s Chair-Stand Test | six-weeks post-operation(T3)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
30s Chair-Stand Test | six-month follow-up
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
40-m Fast-Paced Walk Test | pre-operative session (T1)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
40-m Fast-Paced Walk Test | two-weeks post-operation (T2)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
40-m Fast-Paced Walk Test | six-weeks post-operation(T3)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
40-m Fast-Paced Walk Test | six-month follow-up
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Stair-Climb Test | pre-operative session (T1)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Stair-Climb Test | two-weeks post-operation (T2)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Stair-Climb Test | six-weeks post-operation(T3)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Stair-Climb Test | six-month follow-up
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Timed Up-and-Go Test | pre-operative session (T1)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Timed Up-and-Go Test | two-weeks post-operation (T2)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Timed Up-and-Go Test | six-weeks post-operation(T3)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Timed Up-and-Go Test | six-month follow-up
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
6-min Walk Test | pre-operative session (T1)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
6-min Walk Test | two-weeks post-operation (T2)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
6-min Walk Test | six-weeks post-operation(T3)
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
6-min Walk Test | six-month follow-up
  This test is chosen as recommended by the Osteoarthritis Research Society International Advisory Group (OARSI) for their sensitivity in detecting change in knee functions over time in knee OA patients. Testing and scoring procedures strictly adheres to the standardization and instructions suggested in the OARSI recommendation.
Step Length Asymmetry | pre-operative session (T1)
  Step length is the anterior-posterior (i.e. along the x-axis) distance in millimeters between ankles markers at heel strike. Equal step lengths result in zero step length asymmetry. Step length asymmetry is related to propulsive force generation during paretic walking. In situation where the unaffected leg's step length is longer than the affected leg's step length indicates step length asymmetry. Step length asymmetry is then quantified by using a step length ratio, defined as step length of the (more) affected limb divided by the step length non-affected limb (or less affected limb). This results in a unitless parameter that is essential for comparing inter-subject differences.The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Step Length Asymmetry | two-weeks post-operation (T2)
  Step length is the anterior-posterior (i.e. along the x-axis) distance in millimeters between ankles markers at heel strike. Equal step lengths result in zero step length asymmetry. Step length asymmetry is related to propulsive force generation during paretic walking. In situation where the unaffected leg's step length is longer than the affected leg's step length indicates step length asymmetry. Step length asymmetry is then quantified by using a step length ratio, defined as step length of the (more) affected limb divided by the step length non-affected limb (or less affected limb). This results in a unitless parameter that is essential for comparing inter-subject differences. The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Step Length Asymmetry | six-weeks post-operation(T3)
  Step length is the anterior-posterior (i.e. along the x-axis) distance in millimeters between ankles markers at heel strike. Equal step lengths result in zero step length asymmetry. Step length asymmetry is related to propulsive force generation during paretic walking. In situation where the unaffected leg's step length is longer than the affected leg's step length indicates step length asymmetry. Step length asymmetry is then quantified by using a step length ratio, defined as step length of the (more) affected limb divided by the step length non-affected limb (or less affected limb). This results in a unitless parameter that is essential for comparing inter-subject differences. The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Step Length Asymmetry | six-month follow-up
  Step length is the anterior-posterior (i.e. along the x-axis) distance in millimeters between ankles markers at heel strike. Equal step lengths result in zero step length asymmetry. Step length asymmetry is related to propulsive force generation during paretic walking. In situation where the unaffected leg's step length is longer than the affected leg's step length indicates step length asymmetry. Step length asymmetry is then quantified by using a step length ratio, defined as step length of the (more) affected limb divided by the step length non-affected limb (or less affected limb). This results in a unitless parameter that is essential for comparing inter-subject differences. The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Knee Moment | pre-operative session (T1)
  Knee Moment is a measurement of the medial tibiofemoral contact force. The initial peak knee adduction torque during walking is a strong predictor of the severity and rate of progression of medial compartment knee OA. The KAM is generated by the combination of ground reaction force, which passes medially to the knee joint during walking. It is recorded by two force plates at 1080Hz and 3D kinematic data acquired by the infrared camera system at 120Hz using the VICON Motion System, Oxford, UK. In this particular study, subjects that has been selected to receive 3D bipedal locomotion analysis using the Vicon Optical Motion Capturing system will be assessed under various walking conditions; The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Knee Moment | two-weeks post-operation (T2)
  Knee Moment is a measurement of the medial tibiofemoral contact force. The initial peak knee adduction torque during walking is a strong predictor of the severity and rate of progression of medial compartment knee OA. The KAM is generated by the combination of ground reaction force, which passes medially to the knee joint during walking. It is recorded by two force plates at 1080Hz and 3D kinematic data acquired by the infrared camera system at 120Hz using the VICON Motion System, Oxford, UK. In this particular study, subjects that has been selected to receive 3D bipedal locomotion analysis using the Vicon Optical Motion Capturing system will be assessed under various walking conditions; The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Knee Moment | six-weeks post-operation(T3)
  Knee Moment is a measurement of the medial tibiofemoral contact force. The initial peak knee adduction torque during walking is a strong predictor of the severity and rate of progression of medial compartment knee OA. The KAM is generated by the combination of ground reaction force, which passes medially to the knee joint during walking. It is recorded by two force plates at 1080Hz and 3D kinematic data acquired by the infrared camera system at 120Hz using the VICON Motion System, Oxford, UK. In this particular study, subjects that has been selected to receive 3D bipedal locomotion analysis using the Vicon Optical Motion Capturing system will be assessed under various walking conditions; The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Knee Moment | six-month follow-up
  Knee Moment is a measurement of the medial tibiofemoral contact force. The initial peak knee adduction torque during walking is a strong predictor of the severity and rate of progression of medial compartment knee OA. The KAM is generated by the combination of ground reaction force, which passes medially to the knee joint during walking. It is recorded by two force plates at 1080Hz and 3D kinematic data acquired by the infrared camera system at 120Hz using the VICON Motion System, Oxford, UK. In this particular study, subjects that has been selected to receive 3D bipedal locomotion analysis using the Vicon Optical Motion Capturing system will be assessed under various walking conditions; The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Ground Reaction Force | pre-operative session (T1)
  Ground Reaction Force ( GRF) is a gait variable that has been reported to be closely associated with walking speed, severity of disease and presence of step length asymmetry in knee OA patients. GRF is determined using a frequency threshold of 20Hz, and the resultant force (measured in Newtons) will be normalized using division normalization. It is a common practice for studies evaluating GRF to normalize these forces by linear scaling them to subject's body weight, in order to allow comparison between subjects.The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Ground Reaction Force | two-weeks post-operation (T2)
  Ground Reaction Force ( GRF) is a gait variable that has been reported to be closely associated with walking speed, severity of disease and presence of step length asymmetry in knee OA patients. GRF is determined using a frequency threshold of 20Hz, and the resultant force (measured in Newtons) will be normalized using division normalization. It is a common practice for studies evaluating GRF to normalize these forces by linear scaling them to subject's body weight, in order to allow comparison between subjects.The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Ground Reaction Force | six-weeks post-operation(T3)
  Ground Reaction Force ( GRF) is a gait variable that has been reported to be closely associated with walking speed, severity of disease and presence of step length asymmetry in knee OA patients. GRF is determined using a frequency threshold of 20Hz, and the resultant force (measured in Newtons) will be normalized using division normalization. It is a common practice for studies evaluating GRF to normalize these forces by linear scaling them to subject's body weight, in order to allow comparison between subjects.The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Ground Reaction Force | six-month follow-up
  Ground Reaction Force ( GRF) is a gait variable that has been reported to be closely associated with walking speed, severity of disease and presence of step length asymmetry in knee OA patients. GRF is determined using a frequency threshold of 20Hz, and the resultant force (measured in Newtons) will be normalized using division normalization. It is a common practice for studies evaluating GRF to normalize these forces by linear scaling them to subject's body weight, in order to allow comparison between subjects.The participants will walk in 3 conditions. i: comfortable speed; ii: affected limb accelerated (by 30%) and iii affected limb decelerated (by 30%).
Osteoarthritis Fears and Beliefs Questionnaire (KOBeQ) | pre-operative session (T1)
  Fear avoidance belief will be assessed using self-reported questionnaires, The Knee Osteoarthritis Fears and Beliefs Questionnaire (KOBeQ) Minimum：0 Maximum：99 Higher scores on the KOFBeQ indicate better health status.
Osteoarthritis Fears and Beliefs Questionnaire (KOBeQ) | two-weeks post-operation (T2)
  Fear avoidance belief will be assessed using self-reported questionnaires, The Knee Osteoarthritis Fears and Beliefs Questionnaire (KOBeQ) Minimum：0 Maximum：99 Higher scores on the KOFBeQ indicate better health status.
Osteoarthritis Fears and Beliefs Questionnaire (KOBeQ) | six-weeks post-operation(T3)
  Fear avoidance belief will be assessed using self-reported questionnaires, The Knee Osteoarthritis Fears and Beliefs Questionnaire (KOBeQ) Minimum：0 Maximum：99 Higher scores on the KOFBeQ indicate better health status.
Osteoarthritis Fears and Beliefs Questionnaire (KOBeQ) | six-month follow-up
  Fear avoidance belief will be assessed using self-reported questionnaires, The Knee Osteoarthritis Fears and Beliefs Questionnaire (KOBeQ) Minimum：0 Maximum：99 Higher scores on the KOFBeQ indicate better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No